CLINICAL TRIAL: NCT01040390
Title: Efficacy of Lesser Known Homoeopathic Medicines in Acne Vulgaris - Lappa Arctium
Brief Title: Efficacy of Lappa Arctium (Homoeopathic Medicine) in Treatment of Acne Vulgaris
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Miglani, Anjali (Individual)
Collaborators: Department of Indian Systems of Medicine and Homeopathy (Other)
Responsible Party: Principal Investigator, Dr. Anjali Miglani, Senior Medical Officer, Miglani, Anjali
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Acne-001
Record Dates: First submitted 2009-12-26; First posted 2009-12-29 (Estimated); Last update posted 2012-02-17 (Estimated); Status verified 2012-02

CONDITIONS: Acne Vulgaris
Keywords: Acne Vulgaris; Homoeopathy; Lappa Arctium
MeSH Terms: conditions — Acne Vulgaris

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Lappa Arctium — To start with subjects will be prescribed Lappa Arctium in 6 potency to be taken in form of pills 4 times a day for seven days. Dosage and frequency will be changed, if required, based on the condition of subject and their response according to homoeopathic principles.
  Other Names: Lappa Major

SUMMARY:
Acne is one of the most common skin problems in teenagers and adolescents. There are many lesser known homoeopathic medicines which have been mentioned in the literature for treatment of acne but their potential has not been properly assessed /documented and therefore these medicines don't form a part of many prescriptions. As a part of this study,efficacy of Lappa Arctium will be studied in the treatment of Acne vulgaris

ELIGIBILITY:
Inclusion Criteria:

* Males and females between 12 to 25 years of age
* Presence of inflammatory and non-inflammatory lesions
* Able to follow-up according to protocol
* Patients not taking any medication for treatment of Acne in preceding one month.

Exclusion Criteria:

* Acne Conglobata
* Pregnant or Breast feeding females or females having intention of becoming pregnant
* Significant systemic disease
* Any drug/ alcohol addiction
* History of chronic diseases treated with medications in the preceding month which might affect acne condition and treatment outcome

Ages: 12 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 34 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
percent change in acne lesion counts from the Baseline | 6 months

SECONDARY OUTCOMES:
change in quality of life of subjects | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Anjali Miglani, BHMS, Principal Investigator — Department of Indian Systems of Medicine and Homeopathy
Locations (1):
- Delhi Government Health Centre - Homoeopathic Dispensary - Sector 12, Dwarka, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Miglani A, Manchanda RK. Observational study of Arctium lappa in the treatment of acne vulgaris. Homeopathy. 2014 Jul;103(3):203-7. doi: 10.1016/j.homp.2013.12.002. PMID 24931753